CLINICAL TRIAL: NCT02374606
Title: Accurate Test of Limb Isometric Strength (ATLIS) in ALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Peggy Allred, PT DPT, Research Program Administrator/Neuromuscle Program Manager, Cedars-Sinai Medical Center
Other Study IDs: Pro00038868
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: outcomes measures; strength measurement; disease progression
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A strength measurement device called Accurate Test of Limb Isometric Strength (ATLIS) was developed to precisely and conveniently measure static limb strength in patients with ALS. The investigator will compare ATLIS data with data from the commonly used ALS outcomes measure, the ALS Functional Rating Scale-Revised (ALSFRS-R), as well as an exploratory measure, electrical impedance myography (EIM), in a prospective, longitudinal study. Both outcomes measures will be performed on 100 subjects collected preferably at bi-monthly clinic visits during the study period.

DETAILED DESCRIPTION:
Cedars-Sinai Medical Center will enroll and collect data on 100 subjects. Subjects will ideally be tested every 1 to 4 months according to each patient's site visit schedule. Subjects will be tested at each visit using ATLIS, the ALSFRS-R questionnaire and EIM.

ELIGIBILITY:
Inclusion criteria:

* Subjects 18 years or older diagnosed with clinically possible, laboratory supported probable, probable or clinically definite ALS according to the World Federation of Neurology Revised El Escorial Criteria.
* Capable of providing informed consent and complying with trial procedures.
* Active movement of at least two limbs at the time of study entry
* Intend to routinely attend clinic for neurological care at the clinical site

Exclusion criteria:

* Patients, judged by the site clinical investigator to have medical conditions that may limit their ability to safely exert maximal force using the muscles in their arms and legs will be excluded from this study (e.g. unstable hypertension, significant cardiac disease, significant musculoskeletal disorders, or other medical conditions).
* Patients judged by the site clinical investigator to have significant clinical evidence of unstable medical or psychiatric illness will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ALS
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change in Accurate Test of Limb Isometric Strength (ATLIS) between each visit | every 1 to 4 months according to each patient's site visit schedule
  ATLIS measures isometric strength in 12 muscle groups in the arms and legs. The subject is tested seated in a specially designed chairs with adjustable uprights. The subject's limb is placed in a standard position and maximal force is exerted on the wireless load cell fixed to the upright. Strength data is digitally captured and expressed as a percentage of expected normal.

SECONDARY OUTCOMES:
Change in ALS Functional Rating Scale - Revised (ALSFRS-R) between each visit | every 1 to 4 months according to each patient's site visit schedule
  This questionnaire consists of 12 questions about the subject's ability to function in certain daily activities. Questions are asked in an interview format.

OTHER OUTCOMES:
Exploratory measure: Electrical impedance myography (EIM) data will be compared to ATLIS data. | every 1 to 4 months according to each patient's site visit schedule
  EIM evaluates how electrical current flows through muscle which assists in determining muscle health by measuring electrical current in muscle. 14 muscle groups in the arms and legs will be tested in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Allred, PT DPT, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No